CLINICAL TRIAL: NCT00341263
Title: Study of Maternal and Umbilical Cord Hormone Concentrations in Monochorionic and Dichorionic Pregnancies
Brief Title: Maternal and Umbilical Cord Hormone Concentrations in Twin and Singleton Pregnancies
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999904052; 04-C-N052
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-01

CONDITIONS: Normal Pregnancy
Keywords: Twins; Clinical Research; Endocrinology; Breast Cancer; Biochemical Epidemiology
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Cases - twin pregnancies: Maternal and cord hormones in twins
- Controls - singleton pregnancies: Maternal and cord hormones in singletons

SUMMARY:
This study will examine levels of hormones, such as estrogen and testosterone, in maternal and umbilical cord blood to compare hormones between mothers who are having twins and mothers who are having one baby. It will investigate whether hormone levels in twin versus singleton pregnancies influence the babies' risk of developing breast, prostate, and testicular cancers later in life.

Pregnant women 18 years of age and older who do not have preeclampsia, chronic hypertension, pre-pregnancy or gestational diabetes, thyroid disease, or other major pregnancy complications are eligible for this study. Participants will be recruited from the obstetrics and gynecology practice at the Dartmouth Hitchcock Medical Center in Lebanon, New Hampshire.

Participants will have a blood sample drawn from their arm during their third trimester prenatal visit and again when they are admitted to the hospital for delivery. After the baby is born, a blood sample will be collected from the cut umbilical cord. Information about the pregnancy and delivery will be collected from the mother's medical chart, and information about the baby's size will be obtained from the baby's medical chart.

DETAILED DESCRIPTION:
Epidemiologic data are few but suggest that effects during the prenatal and early life periods may be important in influencing risk of breast, prostate and testicular cancers later in life. In particular, evidence is accumulating for associations with several maternal, perinatal and pregnancy characteristics, including twining. The effect of these factors may be mediated through alterations in hormone levels such as the estrogens and other steroid hormones, to which the embryo and fetus are exposed during pregnancy. Differences in maternal hormone concentrations by maternal and perinatal factors have been noted, though data for most factors are sparse. Furthermore, less is known about the relationships of pregnancy factors to hormones in cord blood, the proximal exposure to the fetus, since most work thus far has been based on hormones in the maternal circulation. In collaboration with investigators at Dartmouth Hitchcock Medical Center, we are collecting maternal and cord blood samples from monochorionic twin, dichorionic twin and singleton pregnancies of similar gestational age to quantify differences in concentrations of several hormones and other pregnancy products. The purpose of the study is to assess the consistency of these data with hypotheses regarding the altered cancer risk daughters of twin pregnancies experience. All data collection is completed. We are currently analyzing the data for development of manuscripts to be submitted for publication.

ELIGIBILITY:
* INCLUSION CRITERIA/EXCLUSION CRITERIA:

Eligible for study are pregnant women 18 years of age and older.

We will try to recruit women who do not have preeclampsia, chronic hypertension, pre-pregnancy or gestational diabetes, thyroid disease or other major pregnancy complications.

CASES:

Eligible women who are pregnant with twins.

CONTROLS (Singletons):

Three control groups will be recruited: two for the mother of twins (one at the third trimester, one at delivery), and one for the twins themselves at delivery.

A singleton pregnancy that meets the eligibility criteria and can be matched to the case pregnancy on gestational age (within 1 week), parity (nulliparous vs. parous) and maternal age (+/- 5 years) will be recruited for study.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Mothers and children treated at Dartmouth Hitchcock Medical Center and Medical School.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2003-11-21; Primary Completion 2009-07-01 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
Hormone concentrations | Pregnancy
  Analysis of maternal and cord blood hormone concentrations inmonochorionic twin, dichorionic twin and singleton pregnancies of similar gestational age--especially with respect to cancer risk.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Troisi, D.Sc., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Darmouth-Hitchcock Medical Center, Hanover, New Hampshire, United States

REFERENCES:
- [Background] Andersson SW, Bengtsson C, Hallberg L, Lapidus L, Niklasson A, Wallgren A, Hulthen L. Cancer risk in Swedish women: the relation to size at birth. Br J Cancer. 2001 May 4;84(9):1193-8. doi: 10.1054/bjoc.2000.1738. PMID 11336470
- [Background] Braun MM, Ahlbom A, Floderus B, Brinton LA, Hoover RN. Effect of twinship on incidence of cancer of the testis, breast, and other sites (Sweden). Cancer Causes Control. 1995 Nov;6(6):519-24. doi: 10.1007/BF00054160. PMID 8580300
- [Background] Buell P. Changing incidence of breast cancer in Japanese-American women. J Natl Cancer Inst. 1973 Nov;51(5):1479-83. doi: 10.1093/jnci/51.5.1479. No abstract available. PMID 4762931